

Protocol ID: IGT\_IGD\_ICE Registry Study\_2019\_10745 Version 2.0

Protocol Title: ICE-Guided Cardiac Interventional Percutaneous Procedures

Project: The Philips ICE Registry

# Author(s):

Project Statistician: Bob Patel, Consulting Statistician

#### **CONFIDENTIALITY STATEMENT**

This document and the information contained herein or attached hereto ("Confidential Material") are confidential and proprietary to ****. This Confidential Material should only be viewed by those individuals or companies that have been given prior authorization to do so by Philips Clinical Affairs.

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Ciassification. | 1 of internal age |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Version: | 1.0 | User Tool ID: | 16.2.6UserTool0025 | Approver: | Kevin Najarian |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 1 of 16 |



# TABLE OF CONTENTS

| 1 | List of Abbreviations | 4 |
|---|---|---|
| 2 | Introduction | 5 |
| 3 | Study Objectives | 5 |
| | 3.1 Primary Objectives | |
| 4 | Investigation Plan | 7 |
| | 4.1 Overall Study Design 4.2 Discussion of Study Design 4.3 Selection of Study Population 4.4 Treatments 4.4.1 Treatment Groups 4.4.2 Randomization 4.5 Control to Minimize Bias | 7<br>8<br>8<br>8 |
| 5 | Efficacy and Safety Variables | 9 |
| | 5.1 Efficacy and Safety Measurements 5.2 Appropriateness of Measurements 5.3 Efficacy Variables 5.3.1 Primary Efficacy Variables 5.3.2 Secondary Efficacy Variables 5.4 Safety Variables | 9<br>9<br>9<br>.10 |
| 6 | Endpoint Definition | .11 |
| 7 | Data Quality Assurance | .11 |
| 8 | Statistical Methods | .12 |
| | 8.1 Sample Size 8.2 General Consideration. 8.2.1 Analysis Population 8.2.2 Handling of Dropouts or Missing Data. | .12<br>.12 |

| Document | ICE VeriSight | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Classification. | 1 of internal use |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 2 of 16 |



| | 8.2.3 Efficacy Subset | 13 |
|----|---------------------------------------------------------|-----|
| | 8.3 Patient Disposition | |
| | 8.4 Demographics and Baseline Characteristics | 13 |
| | 8.5 Compliance | |
| | 8.6 Concomitant Therapy | 13 |
| | 8.7 Efficacy Analysis | 13 |
| | 8.7.1 Primary Efficacy Analysis | 13 |
| | 8.7.2 Secondary Efficacy Analysis | 14 |
| | 8.7.3 Supplementary Efficacy Analysis | 14 |
| | 8.8 Safety Analysis | |
| | 8.9 Subgroup Analysis | 14 |
| | 8.10 Adjustment for Covariates | 14 |
| | 8.11 Multiple Comparison and Multiplicity | 14 |
| 9 | Changes in the Conduct of the Study or Planned Analysis | 15 |
| | 9.1 Changes in the Conduct of the Study | 15 |
| | 9.2 Changes in the Planned Analysis | |
| 10 | References | 15 |
| 11 | Figures | 15 |
| 12 | Tables1 | 5 |
| 10 | Individual Cubicat data Listings | 1 = |
| 13 | Individual Subject data Listings | ı |

| Document | ICE VeriSight | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Classification. | 1 of internal use |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 3 of 16 |



# 1 LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AE | Adverse Event |
| ADE | Adverse Device Effect |
| ANOVA | Analysis of Variance |
| ASD | Atrial Septal Defect |
| CFR | Code of Federal Regulation |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| DDE | Direct Data Entry |
| DICOM | Digital Imaging and Communications in Medicine |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| GCP | Good Clinical Practice |
| ICE | Intracardiac echocardiography |
| ICH | International Conference on Harmonization |
| IRB | Institutional Review Board |
| ISO | International Organization for Standardization |
| PACS | Picture Archiving and Communication System |
| PFO | Patent Foramen Ovale |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis Software |
| TAVR | Transcatheter Aortic Valve Replacement |
| TEE | Transesophageal Echocardiography |
| UADE | Unanticipated Adverse Device Effect |
| USADE | Unanticipated Serious Adverse Device Effect |
| VSD | Ventricular Septal Defect |

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassincation. To inter | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 4 of 16 |



#### 2 INTRODUCTION

Philips Image Guided Therapy Devices has recently developed and received FDA clearance for an intracardiac echocardiography (ICE) catheter (VeriSight/ VeriSight Pro, henceforth referred to as VeriSight in this plan) that has 2D and/or 3D imaging capabilities. These catheters are for use with Philips EPIQ series ultrasound system. VeriSight is intended (indication for use, IFU) for intracardiac and intra-luminal visualization of cardiac and great vessel anatomy and physiology as well as visualization of other devices in the heart. The catheter is intended for imaging guidance only, not treatment delivery, during cardiac interventional percutaneous procedures. A detailed description of VeriSight can be found in the products' IFU.

The current benchmark/ standard of care for image guidance in percutaneous cardiac intervention procedure is transesophageal echocardiography. The major advantage of ICE over TEE is its unique imaging from within the heart, providing shorter image distances to target anatomy or device, and higher resolution. In addition, ICE can be used under conscious sedation thus avoiding the need for esophageal intubation and eliminating the risk for esophageal trauma. Further, ICE may also reduce fluoroscopy exposure to both the patient and the operator.

#### 3 STUDY OBJECTIVES

The overall purpose of this observational multi-center registry is to report real-world performance and safety of VeriSight ultrasound guided ICE imaging in percutaneous cardiac intervention procedures when used in standard clinical practice.

#### 3.1 Primary Objectives

The primary objectives will include the following:

- a) **Technical success** defined by successful delivery of VeriSight to the target intracardiac position and sustained device operation during the procedure
  - Successful device delivery is defined as ability of the VeriSight catheter to reach the target intracardiac anatomical position. Sustained operation of VeriSight is absence of technical complications or procedural delays/ disruption.
- b) **Imaging success** Adequate image quality as determined by the investigator using a Likert scale assessment.

| Document | ICE VeriSight | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassification. | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 5 of 16 |



c) Clinical success - Adequacy of VeriSight imaging for visualization of major cardiac structures, and guiding procedural intervention, and ability to detect/ assess intraprocedural complications.

Clinical success will be measured by ability of VeriSight to adequately guide procedural intervention using the following parameters:

- number of great vessels imaged, number of chambers imaged, including angle of views, axis, and modality
- ii. assessment of key cardiac structures and sizing relevant anatomy
- iii. verification of delivery and/or placement of interventional device (e.g. transeptal puncture devices, closure devices, Left Atrial Appendage Occlusion (LAAO), Patent Foramen Ovale (PFO), Atrial Septal Defect (ASD), Ventricular Septal Defect (VSD), valves (e.g for TAVR), clip devices (e.g. MitraClip), annuloplasty devices (e.g. Cardioband), ablation devices (e.g cryoballoon, RF ablation catheter), leads (leads extraction), etc.)
- iv. assessment of procedural related complication (e.g. cardiac tamponade, pericardial effusion, thrombus) will be documented for each patient based on the procedure type.
- d) **Safety** Device related adverse events periprocedural through discharge or 48 hours post-procedure, whichever is earlier.

# 3.2 Secondary Objectives

Secondary objectives will include the following:

- a) Procedural characterization when using VeriSight measured by
  - v. type of procedure utilizing ICE imaging
  - vi. total procedural room time (door-in to door-out, mins), total procedure time (skin to skin, mins)
  - vii. total fluoroscopy time (mins)
  - viii. total contrast volume used (cc), fluoroscopic dosage (mGy)
  - ix. ability to image from the right side of the heart for a left sided intervention
  - x. TEE usage rate and avoidance of TEE procedure
  - xi. Other imaging modality used during the procedure
  - xii. Change in management from use of VeriSight need for high risk patient and/or procedure management
  - xiii. Duration and type of anesthesia
  - xiv. Freedom from general anesthesia

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 6 of 16 |



- b) Device characterization when using VeriSight based on a scoring scale for the physical attributes of the VeriSight catheter
- c) Physician survey regarding the Philips ICE using a five-point ordinal Likert-type rating scale
- d) Staff survey regarding the Philips ICE using a five-point ordinal Likert-type rating scale

#### 4 INVESTIGATION PLAN

#### 4.1 Overall Study Design

This is a prospective, multi-center, observational, single-arm registry intended to gather real-world data to report VeriSight ICE catheter performance and safety. It will be conducted in the United States under the approval of one or more recognized institutional review boards and in compliance with GCP guidelines defined in ISO:14155, the Declaration of Helsinki, and all applicable federal and local laws and regulations. Only on label uses of the VeriSight ICE catheter will be allowed. No specific claims are being validated during this registry, though data analyzed from this registry are intended to inform future claims regarding the performance and safety of the VeriSight catheter.

Enrolled subjects will be imaged with VeriSight for various types of percutaneous cardiac interventional procedures. Enrolled subjects will be followed until discharge or ≤48 hrs post-procedure. The registry has a planned duration of approximately 24-36 months with interim analysis planned at 100 subjects to conduct safety and performance analysis for data submission toward CE mark application. Therefore, the initial analysis (n=100) may be limited in scope and it is anticipated that enrollment will continue beyond 100 patients. Statistical hypotheses are not intended for this registry and descriptive analysis will be conducted.

Data from all clinical sites are intended to be pooled for analysis. It is possible that sub-analyses may be conducted to demonstrate VeriSight guidance for target intervention types in structural heart and electrophysiology procedures (see section 8.9 for examples).

#### 4.2 Discussion of Study Design

Please refer to section 4.1

#### 4.3 Selection of Study Population

All subjects age 18 and older that are scheduled for and will undergo a planned cardiac interventional percutaneous procedure in which the guidance of ICE is indicated, eligible and willing to sign an informed consent form without meeting any of the exclusion criteria set and

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 7 of 16 |



meeting all the inclusion criteria set forth in the protocol will be included in the population for analyses. Those who sign consent but do not undergo a cardiac procedure utilizing the Philips ICE catheter will be excluded from the analyses (screen failures).

#### 4.4 Treatments

This is a single-arm registry study, so there are no treatments groups

# 4.4.1 Treatment Groups

This is not applicable for the single arm observational study.

#### 4.4.2 Randomization

This is not applicable for the single arm observational study.

#### 4.5 Control to Minimize Bias

The following measures will be taken to minimize and/or avoid bias in this registry:

- a) A multi-center observational registry design is used to help ensure a representative sample of physicians performing the procedure and to provide a reasonable enrollment period.
- b) Sites will have the ability to represent all-comers in various percutaneous cardiac intervention procedures.
- c) Subjects will be screened to confirm study eligibility with defined inclusion/exclusion criteria prior to inclusion. Sites are required to maintain a log of all subjects screened and enrolled for the study.
- d) Data collection requirements and study procedures will be standardized across all sites. All sites will follow the same version of the protocol and eCRFs.
- e) Collection and archiving of image data will be managed adequately to reduce the impact of data loss and error in analysis.
- f) Standardized protocol training will be developed and distributed to all participating sites to ensure data of uniform quality are obtained from all subjects
- g) Regular monitoring will be conducted to verify source data and adherence to the protocol

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassification. To fine | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 8 of 16 |



#### 5 EFFICACY AND SAFETY VARIABLES

The overall purpose of this observational multi-center registry is to report real-world performance (efficacy) and safety of VeriSight ultrasound guided ICE imaging in percutaneous cardiac intervention procedures when used in standard clinical practice.

#### 5.1 Efficacy and Safety Measurements

See Sections 5.3 below.

#### 5.2 Appropriateness of Measurements

Please refer to section 5.3 and 5.4 below .....

# 5.3 Efficacy Variables

#### 5.3.1 Primary Efficacy Variables

- a) **Technical success** defined by successful delivery of VeriSight to the target intracardiac position and sustained device operation during the procedure
  - Successful device delivery is defined as ability of the VeriSight catheter to reach the target intracardiac anatomical position. Sustained operation of VeriSight is absence of technical complications or procedural delays/ disruption.
- b) **Imaging success** Adequate image quality as determined by the investigator using a Likert scale assessment.
- c) Clinical success Adequacy of VeriSight imaging for visualization of major cardiac structures, and guiding procedural intervention, and ability to detect/ assess intraprocedural complications. Clinical success will be measured by ability of VeriSight to adequately guide procedural intervention using the 4 parameters listed below:
  - number of great vessels imaged, number of chambers imaged, including angle of views, axis, and modality
  - assessment of key cardiac structures and sizing relevant anatomy
  - verification of delivery and/or placement of interventional device (e.g. trans septal puncture devices, closure devices (LAAO, PFO, ASD, VSD), valves (e.g for TAVR), clip devices (e.g. mitral clip), annuloplasty devices (e.g. Cardioband), ablation devices (e.g cryoballoon, RF ablation catheter), leads (leads extraction), etc.)

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassification. | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 9 of 16 |



 assessment of procedural related complication (e.g. cardiac tamponade, pericardial effusion, thrombus) will be documented for each patient based on the procedure type.

# 5.3.2 Secondary Efficacy Variables

Secondary analyses will include the following:

- a) Procedural characterization when using VeriSight measured by
  - i. type of procedure utilizing ICE imaging
  - ii. total procedural room time (door-in to door-out, mins), total procedure time (skin to skin, mins)
  - iii. total fluoroscopy time (mins)
  - iv. total contrast volume used (cc), fluoroscopic dosage (mGy)
  - v. ability to image from the right side of the heart for a left sided intervention
  - vi. TEE usage rate and avoidance of TEE procedure
  - vii. Other imaging modality used during the procedure
  - viii. Change in management from use of VeriSight need for high risk patient and/or procedure management
  - ix. Duration and type of anesthesia
  - x. Freedom from general anesthesia
- b) Device characterization when using VeriSight based on a scoring scale for the physical attributes of the VeriSight catheter
- c) Physician survey regarding the Philips ICE using a five-point ordinal Likert-type rating scale
- d) Staff survey regarding the Philips ICE using a five-point ordinal Likert-type rating scale

#### 5.4 Safety Variables

Device related adverse events periprocedural through discharge or 48 hours post-procedure, whichever is earlier.

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Oldoomodilon. | 1 of internal asc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 10 of 16 |



#### **6 ENDPOINT DEFINITION**

The statistical endpoint is a registry trial outcome value that is measured for each subject, for example subject is a success for binary endpoint.

The four key endpoints are:

- 1. Binary end points are yes/no type of measurements.
- 2. Categorical endpoints are categorized measurements such as race, gender. Typical summary measures are frequencies and percentages.
- Continuous endpoints are measured on a numerical scale such as age in years and heights in inches. Typical summary measures are N, mean, median, standard deviation.
- 4. Time to event endpoints.

#### 7 DATA QUALITY ASSURANCE

Each site, both clinical and laboratory (if applicable), should have SOPs for quality management that describe:

- How data will be evaluated for compliance with the protocol, ethical standards, regulatory compliance, and accuracy in relation to source documents.
- The documents to be reviewed (e.g., CRFs, clinic notes, questionnaires, audio or video recordings), who is responsible, and the frequency for reviews.
- Who will be responsible for addressing QA issues (e.g., correcting procedures that are not in compliance with protocol) and QC issues (e.g., correcting errors in data entry).
- Staff training methods and how such training will be tracked.
- If applicable, calibration exercises conducted prior to and during the study to train examiners and maintain acceptable intra- and inter-examiner agreement.

Regular monitoring and an independent audit, if conducted, must be performed according to International Conference on Harmonisation-Good Clinical Practice (ICH GCP).

Each clinical site will perform internal quality management of study conduct, data collection, documentation and completion.

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | 1 of internal asc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 11 of 16 |



Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

#### 8 STATISTICAL METHODS

#### 8.1 Sample Size

A sample size of up to 200 subjects who are scheduled to undergo cardiac interventional percutaneous procedures are planned for the ICE registry and is considered adequate.

No formal statistical hypothesis test is to be performed and the primary and secondary endpoints will also be summarized by descriptive statistics only.

#### 8.2 General Consideration

No formal statistical hypothesis tests are planned. The primarily all data are to be summarized using descriptive statistics only.

The categorical data will be summarized by frequencies and associated percentages. The continuous data will be summarized by appropriates descriptive statistics such as mean, median, mode, standard deviation, and appropriate percentiles.

The response categories, particularly Physician and Staff Survey data, in Likert scales have a rank order, but the intervals between values cannot be presumed equal. Therefore, the mean (and standard deviation) is inappropriate for ordinal data. So, this type of data will be summarized by Percentiles, such as median, proportions, and mode. Display the distribution of data observations in a bar chart.

The exact (Clopper-Pearson) two-sided 95% confidence interval for each of the 3 primary parameters, namely technical success, imaging success, and clinical success will be reported.

The Clopper-Pearson exact method is chosen since it uses exact binomial distribution to provide at least 95% confidence level for the interval for proportions (p) of the three primary efficacy parameters.

#### 8.2.1 Analysis Population

Since registry study is an observational study, no per protocol nor intent-to-treat population analyses is to be performed.

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | 1 of internal asc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 12 of 16 |



## 8.2.2 Handling of Dropouts or Missing Data

Since this is an observational study, only descriptive statistics are reported, and therefore impact of missing data will not be evaluated.

# 8.2.3 Efficacy Subset

No subset of efficacy data summarization is planned. Consequently, subset analyses will not be performed.

## 8.3 Patient Disposition

Enrolled subjects will be followed until discharge or ≤48 hrs post-procedure. A subject is considered to have completed and exited the registry if he or she has completed all phases of the study including the last visit or the last scheduled procedure.

A protocol deviation is defined as an event where the clinical Investigator or site personnel deviate from the registry protocol or study procedures.

#### 8.4 Demographics and Baseline Characteristics

The categorical data will be summarized by frequencies and associated percentages. The continuous data will be summarized by appropriates descriptive statistics such as mean, median, mode, standard deviation, and appropriate percentiles.

#### 8.5 Compliance

This study will be monitored using a risk-based monitoring approach, consistent with the FDA guidance Oversight of Clinical Investigations.

## 8.6 Concomitant Therapy

Not applicable

### 8.7 Efficacy Analysis

The categorical data will be summarized by frequencies and associated percentages. The continuous data will be summarized by appropriates descriptive statistics such as mean, median, mode, standard deviation, and appropriate percentiles.

#### 8.7.1 Primary Efficacy Analysis

The exact (Clopper-Pearson) two-sided 95% confidence interval for each of the 3 primary parameters, namely technical success, imaging success, and clinical success will be reported.

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | 1 of internal asc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 13 of 16 |



The Clopper-Pearson exact method is chosen since it uses exact binomial distribution to provide at least 95% confidence level for the interval for proportions (p) of the three primary efficacy parameters.

# 8.7.2 Secondary Efficacy Analysis

The categorical data such as race, gender, age categorized as old vs young will be summarized by frequencies and associated percentages. The continuous data will be summarized by appropriates descriptive statistics such as mean, median, mode, standard deviation, and appropriate percentiles.

#### 8.7.3 Supplementary Efficacy Analysis

Refer to Section 8.2 above for the details on assessment for Physician and Staff survey data.

# 8.8 Safety Analysis

Due to the nature of this observational real-world registry, a safety oversight/data safety monitoring committee is unnecessary and not planned.

Summary of Adverse Events will consist of reporting Total Number of Events, Subjects with at Least One AE, Subjects with at Least One UADE, Subjects with at Least One UADE, Subjects with at Least One Procedure or Study device related, and Subjects with at Least One ongoing AE.

Incidence of AE with Relationship to study intervention will be summarized by frequencies associated percentages.

#### 8.9 Subgroup Analysis

Subgroup analyses reporting of descriptive statistics for demographic, safety and efficacy parameters as requested may be performed for the procedure types obtained from the registry.

# 8.10 Adjustment for Covariates

Not applicable.

#### 8.11 Multiple Comparison and Multiplicity

Not applicable

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | 1 of internal asc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 14 of 16 |



# 9 CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSIS

# 9.1 Changes in the Conduct of the Study

None

# 9.2 Changes in the Planned Analysis

None

#### 10 REFERENCES

All statistical analyses will be performed using the SAS® software version 9.4

#### 11 FIGURES

Appropriate histogram or bar charts will be reported.

#### 12 TABLES

Statistical summary of analyses will be reported as by appropriate tables which will be provided as a separate document.

# 13 INDIVIDUAL SUBJECT DATA LISTINGS

Data listing supporting statistical tables will be generated.

# **Document Revision History**

| Version | Date | Author | Description of Change | Reason for Change |
|---------|-----------|-----------|-----------------------|-------------------|
| 1.0 | 02SEP2022 | Bob Patel | N/A | Initial release |

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinsation. | 1 of internal acc |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 15 of 16 |



# **Document Approval History**

| Approved by | Role / Function | Signature & Date | |
|---|---|---|---|
| Bob BabaBhai Patel | Project Statistician (SAP author) | Bababhai Patel | Electronically signed by: Bababhai Patel<br>Reason: "I Approve"<br>Date: Sep 2, 2022 19:40 EDT |
| Rashmi Ram, PhD | Project Manager or<br>Business Leader | Rashmi Ram | Electronically signed by: Rashmi Ram<br>Reason: "I Approve"<br>Date: Sep 2. 2022 17:50 MDT |
| Janice Ambers | Clinical Study<br>Manager or Clinical<br>Operations Lead | Forba | Electronically signed by: Janice Ambers<br>Reason: "I Approve"<br>Date: Sep 2, 2022 12:18 PDT |
| Kevin Najarian | Director of<br>Biostatistics | Kevin Najarian | Electronically signed by: Kevin Najarian<br>Reason: "I Approve"<br>Date: Sep 2, 2022 15:25 EDT |
| Sheri Halverson | Associate Director of Clinical Operations | Sheri L. Halverson | Electronically signed by: Sheri Halverson<br>Reason: "I Approve"<br>Date: Sep 2, 2022 19:57 CDT |

| Document | J | Document title: Statistical Analysis Plan | | Classification: | For internal use |
|---|---|---|---|---|---|
| ID: | Registry SAP | | | Olassinoation. | |
| Modified: | 02SEP2022 | | | Author: | Bob Patel |
| Status: | Final | User Tool Version Date: | 29Oct2019 | Page: | 16 of 16 |

# ICE VeriSight Registry SAP

Final Audit Report 2022-09-03

Created: 2022-09-02

By: Janice Ambers (janice.ambers\_1@philips.com)

Status: Signed

Transaction ID: CBJCHBCAABAAW6B-6X-nz4QP1JZC-VyMdKER647Xlv7a

# "ICE VeriSight Registry SAP" History

- Document created by Janice Ambers (janice.ambers\_1@philips.com) 2022-09-02 7:14:44 PM GMT- IP address: 155.190.3.7
- Document emailed to Janice Ambers (janice.ambers\_1@philips.com) for signature 2022-09-02 7:17:30 PM GMT
- Document emailed to kevin.najarian@philips.com for signature 2022-09-02 7:17:30 PM GMT
- Document emailed to Rashmi Ram (rashmi.ram@philips.com) for signature 2022-09-02 7:17:30 PM GMT
- Document emailed to Sheri Halverson (Sheri.Halverson@philips.com) for signature 2022-09-02 7:17:31 PM GMT
- Document emailed to Bababhai Patel (bob.patel@philips.com) for signature 2022-09-02 7:17:31 PM GMT
- Document e-signed by Janice Ambers (janice.ambers\_1@philips.com)

Signing reason: "I Approve"

Signature Date: 2022-09-02 - 7:18:11 PM GMT - Time Source: server- IP address: 155.190.3.7

- Email viewed by kevin.najarian@philips.com 2022-09-02 7:24:17 PM GMT- IP address: 104.47.2.254
- Signer kevin.najarian@philips.com entered name at signing as Kevin Najarian 2022-09-02 7:25:57 PM GMT- IP address: 155.190.19.5
- Document e-signed by Kevin Najarian (kevin.najarian@philips.com)

Signing reason: "I Approve"

Signature Date: 2022-09-02 - 7:25:58 PM GMT - Time Source: server- IP address: 155.190.19.5

Email viewed by Rashmi Ram (rashmi.ram@philips.com) 2022-09-02 - 8:13:51 PM GMT- IP address: 104.47.0.254



Email viewed by Sheri Halverson (Sheri.Halverson@philips.com)

2022-09-02 - 10:07:28 PM GMT- IP address: 104.47.1.254

Email viewed by Bababhai Patel (bob.patel@philips.com)

2022-09-02 - 11:39:29 PM GMT- IP address: 155.190.19.6

Document e-signed by Bababhai Patel (bob.patel@philips.com)

Signing reason: "I Approve"

Signature Date: 2022-09-02 - 11:40:52 PM GMT - Time Source: server- IP address: 155.190.19.6

Document e-signed by Rashmi Ram (rashmi.ram@philips.com)

Signing reason: "I Approve"

Signature Date: 2022-09-02 - 11:50:02 PM GMT - Time Source: server- IP address: 155.190.18.5

Document e-signed by Sheri Halverson (Sheri.Halverson@philips.com)

Signing reason: "I Approve"

Signature Date: 2022-09-03 - 0:57:37 AM GMT - Time Source: server- IP address: 155.190.17.5

Agreement completed.

2022-09-03 - 0:57:37 AM GMT

